CLINICAL TRIAL: NCT02078440
Title: Single Dose Pharmacokinetic Study of CYCLOSET ® 0.8 mg Tablets Following Administration of a Weight-Adjusted Dose in Male and Female Children and Adolescent Type 2 Diabetes Mellitus Subjects VS-PEDS BA-2010-V4
Brief Title: Pharmacokinetic Study of CYCLOSET ® 0.8 mg Tablets in Children and Adolescent Type 2 Diabetes Mellitus Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VeroScience (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VS-PEDS BA-2010
Record Dates: First submitted 2014-01-23; First posted 2014-03-05 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Children; Adolescents; Bioavailability; Cycloset; Bromocriptine Mesylate
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Bromocriptine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bromocriptine mesylate (Cycloset) (Other): Bromocriptine mesylate (Cycloset)
  Interventions: Drug: Bromocriptine mesylate

INTERVENTIONS:
Drug: Bromocriptine mesylate — Cycloset (bromocriptine mesylate quick release) 0.8 mg tablets, weight adjusted 1.6 mg- 4.8 mg
  Other Names: Cycloset; Bromocriptine-QR; BQR

SUMMARY:
The objective of this study is to evaluate the relative bioavailability, and the rate and extent of absorption of bromocriptine in male and female children and adolescent Type 2 Diabetes Mellitus patients, aged 10 to less than 18, under fed conditions.

It is undetermined if the pharmacokinetic profile of bromocriptine-QR in type 2 diabetes children aged 10- to less than 18 years differs appreciably from that in healthy adults. Bromocriptine is extensively metabolized by the liver (namely CYP3A4). Studies in children have demonstrated little difference in clearance among children over 10 years of age compared to adults (Blanco et al, 2000). However, differences in blood volumes or other factors may impart differences that could affect the pharmacokinetic properties of bromocriptine-QR. Therefore, this study will assess the pharmacokinetics in children aged 10-to less than 18 years who have type 2 diabetes. After describing the profile of bromocriptine-quick release in this patient population, a follow on study will be conducted to evaluate its safety and efficacy in treating children and adolescents who have type 2 diabetes.

The pharmacokinetic profile of bromocriptine will be determined following the administration of a single, weight-adjusted dose of CYCLOSET (bromocriptine mesylate) tablets. The study will be a single period, bioavailability study in 30 patients. The study duration will be 3 days.

DETAILED DESCRIPTION:
The study is a multi-center, single dose, open-label, 1-period design. Thirty (30) patients will be enrolled in the study and at least twenty-four (24) patients are expected to complete the study.

Male and female patients with confirmed Type 2 Diabetes, non-or ex-smokers, aged 10 to less than 18 years will be selected according to the inclusion and exclusion criteria.

Patients will be admitted to the clinical site at least 10 hours prior to drug administration which will occur within 2 hours of waking on the morning of Day 2.

Ondansetron hydrochloride will be administered orally, approximately 6 hours before the dosing time of Cycloset (bromocriptine mesylate). Subjects weighing 50 to 60 kg will receive 6mg ondansetron hydrochloride (liquid 7.5 ml) and subjects weighing ≥60 kg will receive ondansetron hydrochloride 8 mg (liquid 10 ml).

A single, weight-adjusted dose of CYCLOSET (bromocriptine mesylate), of approximately 0.048 mg/kg, will be administered orally with 240 mL of water in the morning, after a 10-hour overnight fast, and thirty minutes after the start of a standardized breakfast that meets American Diabetes Association diet recommendations.

On day 2, after a supervised overnight fast, the patients will be awakened, vital signs (blood pressure, pulse rate and body temperature) will be measured and the first blood sample (T= 0) will be collected.

Seventeen (17) blood samples will be collected for pharmacokinetic sampling at 0.25, 0.50, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24 and 36 hours post drug administration.

Finger sticks for blood glucose levels will be obtained every hour for the first 4 hours following administration of bromocriptine mesylate, and then additionally as deemed necessary by the study physician.

Safety will be evaluated through the assessment of adverse events and laboratory tests and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Availability for entire study and willingness to adhere to protocol requirements as evidenced by (ICF) duly read, signed and dated by the patient and responsible parent or guardian
* Positive diagnosis of T2DM according to ADA criteria. There is no requirement for time since diagnosis as long as ADA guidelines have been followed.
* Aged at least 10 years but less than 18 years at time of enrollment
* BMI greater than 80th percentile for age and sex and body weight equal to or greater than 50 kg
* Clinical laboratory values within the laboratory's stated normal range - if not within this range, they must be without any clinical significance
* Healthy according to the medical history, laboratory results and physical examination
* Non- or ex-smokers (defined as someone who completely stopped smoking for at least 30 days before day 1 of this study).

Exclusion Criteria:

* Evidence to indicate a diagnosis of Type 1 diabetes
* Body weight less than 50 kilograms
* Systolic blood pressure lower than 115mmHg or diastolic blood pressure lower than 68 mmHg
* Significant history of hypersensitivity to bromocriptine mesylate, ondansetron, other ergot alkaloids or any related products, including excipients of the formulation as well as severe hypersensitivity reactions (like angioedema) to any drugs
* Presence of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects
* Serum aspartate aminotransferase (AST) greater than 3X ULN, and/or serum alanine aminotransferase (ALT) greater than 3X ULN, and/or serum total bilirubin greater than 2.0 mg/dL.
* Calculated glomerular filtration rate less than 80 mL/min based on the Schwartz Formula
* Presence or history of uncontrolled hypertension: systolic pressure greater than 145 mmHg and/or diastolic pressure greater than 95 mmHg, hypertensive disorders of pregnancy, hypertension post-partum and in the puerperium
* History of surgery that may affect drug bioavailability, including but not limited to cholecystectomy
* Presence of significant cardiovascular, pulmonary, hematologic, neurologic, psychiatric, endocrine, immunologic or dermatologic disease
* Symptoms and/or history of serious psychiatric or psychotic disorders
* Presence of significant heart disease or disorder according to ECG
* Presence of malignancy, particularly pituitary gland malignancy and prolactinoma
* Presence or history of migraine headache or syncope
* Pregnant according to a positive serum pregnancy test or lactating
* Females less then four months post-partum
* Current history of illicit drug dependency, use or alcohol abuse (greater than 3 units of alcohol per day, intake of excessive alcohol, acute or chronic).
* Use of drugs for the treatment of ADD and ADHD
* Inhaled corticosteroid use other than as a rescue treatment in case of asthma attack. Use of oral glucocorticoids. Use of oral steroids within the 60 days prior to study entry.
* Any clinically significant illness in the previous 28 days before day 1 of this study
* Use of any cytochrome P450 (CYP) 3A4 enzyme-modifying drugs, including strong inhibitors of CYP 3A4 enzymes and strong inducers of CYP3A4 enzymes (such as barbiturates, carbamazepine, phenytoin and rifampin), in the previous 28 days before Day 1 of this study
* Participation in another clinical trial or donation of 50 mL or more of blood in the previous 42 days before day 1 of this study
* Donation of 500 mL or more of blood in the previous 56 days before Day 1 of this study, as well as donation in excess of 900 mL of blood over the previous 20 weeks
* Positive urine screening of drugs of abuse
* Positive results to HIV, HBsAg or anti-HCV tests

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2014-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | Thirty-six hours
  The pharmacokinetic parameters of interest will be Cmax, AUCT and AUC∞ and Tmax. Other parameters including AUCT/∞, Kel, T½el,CL/F, and Vd, will be provided for information purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Bindu Chamarthi, MD MMSc, Study Director — VeroScience
Locations (5):
- United States (5):
  - Hope Research Institute, Llc, Phoenix, Arizona
  - Yale Center for Clinical Investigation, New Haven, Connecticut
  - Columbus Clinical Services LLC, Miami, Florida
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Children's Hosptial of Philadelphia, Philadelphia, Pennsylvania